CLINICAL TRIAL: NCT05353647
Title: A Multi-Center, Phase 2 Gene Transfer Study Inducing Fetal Hemoglobin in Sickle Cell (GRASP, BMT CTN 2001)
Brief Title: A Gene Transfer Study Inducing Fetal Hemoglobin in Sickle Cell Disease (GRASP, BMT CTN 2001)
Acronym: GRASP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Williams (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other); Genetix Biotherapeutics Inc. (Industry); Blood and Marrow Transplant Clinical Trials Network (Network)
Responsible Party: Sponsor-Investigator, David Williams, Chief - Division of Hematology/Oncology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00038082; 1OT2HL154815 (NIH); CLIN2-12031 (Other Grant/Funding Number: California Institute for Regenerative Medicine)
Record Dates: First submitted 2022-04-21; First posted 2022-04-29 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: gene therapy; lentivirus vector; BCL11A; fetal hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, multi-center, phase 2, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Open-label, non-randomized, single arm study of a single infusion of autologous CD34+ HSC cells transduced with the lentiviral vector containing a shRNA targeting BCL11a.
  Interventions: Biological: Autologous CD34+ HSC cells transduced with the lentiviral vector containing a shRNA targeting BCL11a

INTERVENTIONS:
Biological: Autologous CD34+ HSC cells transduced with the lentiviral vector containing a shRNA targeting BCL11a — A single infusion of autologous CD34+ HSC cells transduced with the lentiviral vector containing a shRNA targeting BCL11a

SUMMARY:
A promising approach for the treatment of genetic diseases is called gene therapy. Gene therapy is a relatively new field of medicine in which genetic material (mostly DNA) in the patient is changed to treat his or her own disease. In gene therapy, we introduce new genetic material in order to fix or replace the patient's disease gene, with the goal of curing the disease. The procedure is similar to a bone marrow transplant, in that the patient's malfunctioning blood stem cells are reduced or eliminated using chemotherapy, but it is different because instead of using a different person's (donor) blood stem cells for the transplant, the patient's own blood stem cells are given back after the new genetic material has been introduced into those cells. This approach has the advantage of eliminating any risk of graft versus host disease (GVHD), reducing the risk of graft rejection, and may also allow less chemotherapy to be utilized for the conditioning portion of the transplant procedure. To introduce new genetic material into the patient's own blood stem cells we use a modified version of a virus (called a 'vector') that efficiently inserts the "correcting" genetic material into the cells. The vector is a specialized biological medicine that has been formulated for use in human beings.

Fetal hemoglobin (HbF) is a healthy, non-sickling kind of hemoglobin. The investigators have discovered a gene that is very important in controlling the amount of HbF. Decreasing the expression of this gene in sickle cell patients could increase the amount of fetal hemoglobin while simultaneously reducing the amount of sickle hemoglobin in their blood, specifically the amount in red blood cells where sickle hemoglobin causes damage to the cell, and therefore potentially cure or significantly improve the condition. The gene we are targeting for change in this study that controls the level of fetal hemoglobin is called BCL11A.

In summary, the advantages of a gene therapy approach include: 1) it can be used even if the patient does not have a matched donor available; 2) it may allow a reduction in the amount of chemotherapy required to prepare the patient for the transplant; and 3) it will avoid certain strong medicines often required to prevent and treat GVHD and rejection. Our lab studies with normal mice, mice that have a form of SCD, and with cells from the bone marrow of SCD patients who have donated bone marrow for research purposes show this approach is very effective in reducing the amount of sickle hemoglobin in red cells. Our pilot trial testing this approach in 10 patients with SCD has shown that the treatment has not caused any unexpected safety problems, and that it increases HbF within the red blood cells. Our goal is to continue to test whether this approach is safe, and whether using gene therapy to change the expression of BCL11A will lead to decreased episodes of vaso-occlusive crisis pain in people with SCD.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center, phase 2 study involving a single infusion of autologous bone marrow derived CD34+ HSC cells transduced with the lentiviral vector containing a short-hairpin RNA targeting BCL11a. 25 patients ages 13 to 40 will be enrolled at sites across the US.

The main goal of this study is to determine whether the treatment will lead to a complete absence of severe vaso-occlusive events (VOEs) in patients with severe SCD.

After meeting eligibility criteria for the study, patients will receive blood transfusions for a period of at least 3 months prior to hematopoietic stem cell collection, with a goal of achieving a HbS level ≤ 30% by the time of mobilization. Patients will then undergo peripheral stem cell mobilization and have their cells collected by apheresis. The collected cells of each subject will be split into 2 portions; one portion for transduction with the lentiviral vector, and one portion set aside as a back-up product in the event a rescue treatment is needed. Patients may undergo multiple rounds of collection if sufficient numbers of cells are not obtained with the first collection. Transduction will be carried out on the selected CD34+ cells and transduced cells will be cryopreserved.

Patients will undergo standard work-up for autologous bone marrow transplantation prior to proceeding with conditioning and infusion of gene-modified cells. Patients will receive myeloablative conditioning with busulfan administered on days -5 to -2, prior to infusion of transduced cells. The transduced cells will be infused intravenously over 30-45 minutes after standard pre-hydration and premedication according to institutional guidelines.

Patients will be followed for 24 months post-infusion of gene modified cells.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of sickle cell disease with genotype HbSS or HbS/β0 thalassemia.
2. Between the age of 13-40 years.
3. Clinically severe disease, defined as at least 4 vaso-occlusive events (VOEs) within the past 24 months prior to consent.
4. Adequate hematologic parameters (regardless of therapy) including white blood cell (WBC) count within the range of 2.5 - 25.0 x 10^9 /L, hemoglobin within the range of 5 - 11 g/dL, and platelet count above 150 x 10^9 /L
5. Adequate organ function and performance status:

   1. Karnofsky/Lansky performance status ≥80%.
   2. Serum creatinine </= 1.5 times the upper limit of normal for age, and calculated creatinine clearance or GFR >/= 60 mL/min/1.73 m2.
   3. Persistent aspartate transaminase, alanine transaminase, or direct bilirubin value <3× the upper limit of normal (ULN).
   4. DLCO, FEV1, and FVC >50% of predicted
   5. Left ventricular ejection fraction >40% or shortening fraction >25%
6. No HLA-genotypically identical related bone marrow donor available.
7. Parental/guardian/patient signed informed consent.

Exclusion Criteria: Subjects who have:

1. Concomitant condition or illness including: ongoing or active infection, active malignancy, major surgery in the past 30 days, medical/psychiatric illness/social situations that would limit compliance with study requirements as determined by the treating physician.
2. Receiving a chronic transfusion regimen for primary or secondary stroke prophylaxis. (Note: patients with a history of abnormal TCD who have transitioned from transfusions to hydroxyurea for stroke prophylaxis are also not eligible for the study.)
3. Patients with history of abnormal TCD (measured with a timed average maximum mean velocity of ≥200 cm/second in the terminal portion of the internal carotid or proximal portion of middle cerebral artery or if the imaging TCD method is used, >185 cm/second plus evidence of intracranial vasculopathy) who were ever on transfusions and subsequently transitioned to hydroxyurea.
4. History of overt stroke or any neurologic event lasting >24 hours. (Note: patients with imaging evidence of silent stroke but not on a chronic transfusion regimen are not excluded.)
5. Isolated recurrent priapism unresponsive to medical and surgical therapies in the absence of other qualifying VOE complications that meet inclusion criteria.
6. Contraindication to administration of conditioning medication (busulfan)
7. Prior allogeneic hematopoietic stem cell transplant
8. Known myelodysplasia of the bone marrow or abnormal bone marrow cytogenetics
9. Severe cerebral vasculopathy
10. Liver MRI (≤ 180 days prior to initiation of BU conditioning) to document hepatic iron content is required for participants who have received ≥20 packed red blood cell transfusions (cumulative); participants who have hepatic iron content ≥ 9 mg Fe/g liver dry weight by liver MRI must have a liver biopsy and histological examination/documentation of the absence of cirrhosis, bridging fibrosis, and active hepatitis (≤ 180 days prior to initiation of transplant conditioning); the absence of bridging fibrosis will be determined using the histological grading and staging scale as described by Ishak and colleagues (1995) as described in the Manual of Operations (MOO);
11. Evidence of HIV infection, HTLV infection, active hepatitis B infection or active hepatitis C infection.
12. Known acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on prior biopsy
13. Receipt of an investigational study drug or procedure within 90 days of study enrollment
14. Either or both of the following findings on screening bone marrow aspirate/biopsy: a) diagnosis of myelodysplastic syndrome (MDS) based on morphology and/or cytogenetics (based on WHO definitions) OR b) pathogenic mutation in any gene on the Rapid Heme Panel (RHP), a next-generation sequencing clinical assay for gene mutations associated with hematologic malignancies performed at Brigham and Women's Hospital.
15. Pregnancy or breastfeeding
16. Presence of a genetically-determined hypercoagulable state or personal history of prior VTE (deep vein thrombosis or pulmonary embolism) that would represent a contraindication to proceed with central line placement and study events.

The Phase 2 trial is not enrolling patients who reside outside the US at this time.

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of VOEs by Month 24 post-infusion | Month 6 to Month 24 post-infusion of gene modified cells
  Each patient will be classified as either a success or a failure (binary endpoint). Success is defined as a complete absence of severe VOEs (defining VOE as a painful event or ACS with no medically determined cause other than a vaso-occlusion, requiring a ≥24-hour hospital or emergency room (ER) observation unit visit or at least 2 visits to a day unit or ER over 72 hours with both visits requiring parenteral opioids) in the period from Month 6 to Month 24 after gene therapy. Patients with one or more severe VOEs from Month 6 to Month 24 after gene therapy, or who experience engraftment failure, or who initiate disease modifying agent(s) for prevention or management of severe VOEs, or who have less than 24 months of follow-up post-infusion, will be classified as 'failures'. For the purpose of this primary endpoint analysis, the first 6 months after infusion of the gene therapy product will be excluded from the VOE observation period.

SECONDARY OUTCOMES:
Hemoglobin Function | Baseline through Month 24 post-infusion of gene modified cells
  Each patient will be classified in terms of hemoglobin function, either sufficient or insufficient (binary endpoint). Sufficient Hb function is defined as either (total Hb of at least 10 g/dL or increase of > 2 g/dL over baseline) and (total HbF > 20% with > 60% F cells). Each of these factors will be measured at Month 9, 12, 15, 18 and 24 post-infusion of gene modified cells. For each factor, the average value across the available time points (minimum of two required) will be utilized to determine if the function criteria have been met, to calculate the binary endpoint
Hemolysis | up to 18 months post-infusion of gene modified cells
  Values of absolute reticulocyte count [units]
Hemolysis | up to 18 months post-infusion of gene modified cells
  Values of lactate dehydrogenase [units]
Hemolysis | up to 18 months post-infusion of gene modified cells
  Values of bilirubin [units]
Toxicities and Adverse Events | Study enrollment through Month 24 post-infusion of gene modified cells
  Adverse events (AEs) grade ≥2 according to CTCAE Version 5 that are related or possibly related to the study procedure, from study enrollment through 24 months.
Percentage change in the annualized number of VOEs | 24 months prior to consent and 6 months to 24 months post-infusion of gene modified cells
  For each evaluable patient (pt), % change in annualized # of severe VOEs will be calculated as:
  (B - A) / A * 100%. A=annualized number of severe VOEs over the 24-month period prior to consent; B=annualized number of severe VOEs from Months 6-24 after gene therapy. For A, annualized # of severe VOEs = [(# of severe VOEs) / 2 years]. For B, annualized number of severe VOEs = [(# of severe VOEs) / (# of years of observation from Month 6-24 post-infusion)].
  For evaluable pts who are lost to follow-up/die/withdraw between Month 6-24, B will be imputed based on the severe VOE rate observed during the time period from Month 6 until the time the pt is lost/dies/withdraws. The minimum length of the VOE observation period required for imputing the annualized VOE rate will be from Month 6 to Month 18 post-infusion. Example: 2 VOEs Month 6-18 (0.167/month) then lost to follow-up; the imputed # of VOEs Month 6-24 equals 3, and annualized B=2.
Occurrence of VOEs by Month 18 post-infusion | Month 6 to Month 18 post-infusion of gene modified cells
  Each patient will be classified as either a complete reduction or not a complete reduction in the number of severe VOEs (binary endpoint). A complete reduction is defined as having no severe VOEs (defining VOE as ACS or VOC requiring parenteral opioids) in a VOE observation period from Month 6 to Month 18 after gene therapy, as compared to the 24 months prior to consent. For the purpose of analysis, the initial 6 months after infusion will be excluded from the VOE observation period.

CONTACTS AND LOCATIONS:
Overall Officials: David Williams, Principal Investigator — Boston Children's Hospital
Locations (9):
- United States (9):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UC Davis Medical Center, Sacramento, California
  - Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No